CLINICAL TRIAL: NCT02471443
Title: Laparoscopic Surgery for Severe Recto-vaginal Endometriosis: A Prospective Cohort Study
Brief Title: Laparoscopic Surgery for Severe Recto-vaginal Endometriosis
Status: Recruiting | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mr Andrew Kent, Consultant Gynaecologist, Royal Surrey County Hospital NHS Foundation Trust
Other Study IDs: 15DEV0009
Record Dates: First submitted 2015-06-06; First posted 2015-06-15 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Endometriosis Rectovaginal Septum
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgery for severe endometriosis: Consecutive patients undergoing excisional surgery for severe endometriosis with bowel involvement
  Interventions: Procedure: Surgery for severe endometriosis

INTERVENTIONS:
Procedure: Surgery for severe endometriosis — Consecutive patients undergoing excisional surgery for severe endometriosis with bowel involvement

SUMMARY:
To determine the quality of life following the radical excision of recto-vaginal endometriosis.

DETAILED DESCRIPTION:
Patients undergoing surgery for severe endometriosis with bowel involvement were asked to complete pre-operative and post operative questionnaires at 2, 6 and 12 months, then 5, 10, 15, 20 and 25 years post operatively.

Quality of life measured using the EHP-30 and EQ-5D questionnaires. Bowel symptoms were measured using GIQLI. Dysmenorrhoea, dyspareunia, dyschezia and chronic pain were measured using a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing planned surgery for severe endometriosis with bowel involvement.

Exclusion Criteria:

* Patients who declined to complete questionnaires for whatever reason and/or have their anonymous data analysed.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who underwent surgery for endometriosis with bowel involvement.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2004-05; Primary Completion 2025-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life measured using the Endometriosis Health Profile 30 (EHP-30) and EuroQol-5 dimension (EQ-5D) questionnaires. | 1 year post operative
  Recruitment is continuous
Bowel symptoms measured using the Gastro-intestinal Quality of Life Index (GIQLI). | 1 year post operative
  Recruitment is continuous
Dysmenorrhoea measured using a visual analogue scale (VAS). | 1 year post operative
  Recruitment is continuous
Dyspareunia measured using a visual analogue scale (VAS). | 1 year post operative
  Recruitment is continuous
Dyschezia measured using a visual analogue scale (VAS). | 1 year post operative
  Recruitment is continuous
Chronic pain measured using a visual analogue scale (VAS). | 1 year post operative
  Recruitment is continuous

SECONDARY OUTCOMES:
Quality of life measured using the EHP-30 and EQ-5D questionnaires. | 2 months, 6 months, 5 years, 10 years, 15 years, 20 years, 25 years follow up post operative
Bowel symptoms were measured using GIQLI. | 2 months, 6 months, 5 years, 10 years, 15 years, 20 years, 25 years follow up post operative
Dysmenorrhoea measured using a visual analogue scale. | 2 months, 6 months, 5 years, 10 years, 15 years, 20 years, 25 years follow up post operative
Dyspareunia measured using a visual analogue scale. | 2 months, 6 months, 5 years, 10 years, 15 years, 20 years, 25 years follow up post operative
Dyschezia measured using a visual analogue scale. | 2 months, 6 months, 5 years, 10 years, 15 years, 20 years, 25 years follow up post operative
Chronic pain measured using a visual analogue scale. | 2 months, 6 months, 5 years, 10 years, 15 years, 20 years, 25 years follow up post operative

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kent, TD MD FRCOG, Principal Investigator — Royal Surrey County Hospital/Nuffield Health Guildford Hospital
Locations (1):
- Royal Surrey County Hospital NHS Trust, Guildford, Surrey, United Kingdom